CLINICAL TRIAL: NCT02433938
Title: Role of Tibial Nerve Stimulation for Enhanced Postoperative Recovery After Colorectal Surgery
Acronym: TiRex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Jacopo Martellucci, MD, PhD, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: jm-001
Record Dates: First submitted 2015-04-09; First posted 2015-05-05 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Ileus; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Underwent tibial nerve stimulation (Experimental): Patients that underwent standard postoperative protocol + tibial nerve stimulation for 3 days
  Interventions: Procedure: Tibial nerve stimulation
- Did not undergo tibial nerve stimulation (Sham Comparator): Patients that underwent standard postoperative protocol + sham tibial nerve stimulation (standard postoperative protocol+sham tns)
  Interventions: Procedure: Sham tibial nerve stimulation

INTERVENTIONS:
Procedure: Tibial nerve stimulation — patients underwent a three days postoperative transcutaneous tibial nerve stimulation
  Arms: Underwent tibial nerve stimulation
Procedure: Sham tibial nerve stimulation — patients did not undergo a postoperative transcutaneous tibial nerve stimulation
  Arms: Did not undergo tibial nerve stimulation

SUMMARY:
Aim of the study is to evaluate the role of postoperative tibial nerve stimulation in the enhancement of the recovery of bowel function and in shortening the hospital stay.

DETAILED DESCRIPTION:
Patients were randomized in two groups. The first group underwent a three days postoperative transcutaneous tibial nerve stimulation. The second group underwent a sham stimulation. Aim of the study is to evaluate the role of tibial nerve stimulation in the postoperative recovery after colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients that underwent colorectal surgery

Exclusion Criteria:

* Severe comorbidities
* Postoperative or intraoperative complications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
bowel function recovery (Time to first bowel movement or flatus) | 7 days
  Time to first bowel movement or flatus

SECONDARY OUTCOMES:
Length of postoperative hospital stay | 30 days
  Length of postoperative hospital stay
Post-operative vomiting (episodes of vomiting) | 30 days
  Episodes of vomiting
Use of NG Tubes (Nasogastric tube (re)insertions) | 30 days
  Nasogastric tube (re)insertions

CONTACTS AND LOCATIONS:
Overall Officials: Jacopo Martellucci, MD, PhD, Study Chair — University of Florence